CLINICAL TRIAL: NCT02792790
Title: Carpal Tunnel Syndrome and Amyloid Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mazen Hanna MD, Prinicipal Investigator, The Cleveland Clinic
Other Study IDs: 16-158
Record Dates: First submitted 2016-04-20; First posted 2016-06-08 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Amyloidosis; Cardiomyopathy; Transthyretin Amyloidosis; Senile Systemic Amyloidosis; Carpal Tunnel Syndrome
Keywords: Amyloidosis; Carpal tunnel syndrome
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies; Amyloidosis, Hereditary, Transthyretin-Related; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be stored in Cleveland Clinic to be used for the future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with carpal tunnel syndrome.: Patients undergoing carpal tunnel release surgery.

SUMMARY:
The investigators will prospectively evaluate tissue samples obtained from patients undergoing carpal tunnel release surgery for amyloid in the soft tissue that is removed. Patients who have tissue that stains positive for amyloid will undergo cardiac testing to look for evidence of cardiac involvement.

DETAILED DESCRIPTION:
Since the 1970s, the connection between amyloidosis and carpal tunnel syndrome has been described, with tenosynovial tissue staining positive for amyloid fibril deposition. Up to 30% of patients in prior studies with idiopathic carpal tunnel syndrome have biopsy tissue that stains positive for amyloid deposition. However, the prevalence of cardiac involvement at the time of carpal tunnel syndrome surgery has not been established. Furthermore, the role of TTR kinetic stability in the disease progression of amyloidosis is unclear.

Diagnosing TTR amyloidosis at the time of carpal tunnel involvement could lead to an earlier identification of the disease at a stage where the cardiomyopathy may be occult or less advanced. In addition, abnormal TTR kinetics may even precede tissue deposition in the flexor tendon retinaculum. As several emerging pharmacological strategies are in development that may slow or even halt TTR amyloidosis, earlier diagnosis is advantageous. Identification and implementation of therapy for prevention or early disease treatment may alter the natural history of this progressive systemic disease.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 50 years of age
* Females ≥ 60 years of age
* Undergoing carpal tunnel release surgery (adequate symptoms are not responding to conservative management requiring surgery)
* Able to consent
* Underwent carpal tunnel surgery and biopsy within last 30 days, if the study was discussed prior to surgery by one of the study physicians.

Exclusion Criteria:

* Secondary CTS (Hemodialysis, rheumatoid arthritis, trauma)
* Known diagnosis of amyloidosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing carpal tunnel release surgery for idiopathic carpal tunnel syndrome not responding conservative and medical management.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of transthyretin (TTR) amyloidosis in patients undergoing carpal tunnel release surgery | Biopsy completed on day of surgery
  Identify the incidence of TTR amyloid deposits in the soft tissue of patients undergoing carpal tunnel surgery for idiopathic carpal tunnel syndrome
Cardiac progression of transthyretin (TTR) amyloidosis in carpal tunnel biopsy-positive patients | 4 years from baseline cardiac assessment.
  Assess the progression of cardiac disease in patients with TTR deposits found in soft tissue removed at the time of carpal tunnel surgery

SECONDARY OUTCOMES:
Prevalence of abnormal transthyretin (TTR) kinetics in patients undergoing carpal tunnel surgery | One-time kinetics test for biopsy-negative patients; baseline kinetics and annually for 4 years in biopsy-positive patients
  Identify the prevalence of abnormal TTR kinetics in patients undergoing carpal tunnel surgery for idiopathic carpal tunnel syndrome (develop a new test that aids identification of misfolded TTR intermediates that is more specific and sensitive to diagnosis this disease in the blood or tissue)
Early transthyretin (TTR) amyloid cardiomyopathy identification in carpal tunnel biopsy-positive patients | Baseline and annual testing for 4 years in biopsy-positive patients
  Investigate whether early TTR cardiomyopathy can be identified in patients who have TTR amyloid deposits identified in the soft tissue removed at the time of carpal tunnel surgery using cardiac biomarkers, echocardiography with strain, and nuclear bone scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Hanna, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Lutheran Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sperry BW, Reyes BA, Ikram A, Donnelly JP, Phelan D, Jaber WA, Shapiro D, Evans PJ, Maschke S, Kilpatrick SE, Tan CD, Rodriguez ER, Monteiro C, Tang WHW, Kelly JW, Seitz WH Jr, Hanna M. Tenosynovial and Cardiac Amyloidosis in Patients Undergoing Carpal Tunnel Release. J Am Coll Cardiol. 2018 Oct 23;72(17):2040-2050. doi: 10.1016/j.jacc.2018.07.092. PMID 30336828